CLINICAL TRIAL: NCT00849875
Title: Study of GSK2132231A Antigen-Specific Cancer Immunotherapeutic in Association With Chemotherapy in Patients With Unresectable and Progressive Metastatic Cutaneous Melanoma
Brief Title: A Study of Safety and Clinical Activity of Immunotherapy Plus Chemotherapy in Metastatic Melanoma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early end of trial notification after termination of long term follow up due to lack of scientific justification to continue collect information.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111714
Record Dates: First submitted 2009-02-02; First posted 2009-02-24 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Melanoma
Keywords: ASCI; Dacarbazine; Cancer immunotherapeutic; MAGE-A3; Malignant melanoma
MeSH Terms: conditions — Melanoma | interventions — Dacarbazine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group A (Experimental): All patients are to receive the same treatment consisting of 24 injections of the immunotherapeutic GSK2132231A combined with a course of 8 cycles of dacarbazine given at the beginning of the treatment
  Interventions: Biological: Immunotherapeutic GSK2132231A; Drug: Dacarbazine

INTERVENTIONS:
Biological: Immunotherapeutic GSK2132231A — Intramuscular administration
Drug: Dacarbazine — Intravenous administration Chemotherapy
  Other Names: DTIC; Imidazole Carboxamide; DTIC-Dome

SUMMARY:
The purpose of this clinical trial is to find out how successfully, patients with progressive metastatic cutaneous melanoma, are able to develop an immune response to injections with the immunotherapeutic product GSK1572932A when given in combination with dacarbazine and evaluate the safety of this combination.

DETAILED DESCRIPTION:
This Protocol Posting has been updated following amendment 3, dated 16 October 2009. The sections impacted are :

* Enrollment, number of subjects
* Outcome measures
* Exclusion criteria

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient with histologically proven, measurable metastatic cutaneous melanoma
2. Written informed consent has been obtained from the patient before the performance of any protocol-specific procedure.
3. Patient is >= 18 years of age at the time of signature of the Informed Consent.
4. The patient's tumor shows expression of MAGE-A3 antigen, detected by Reverse-Transcription Polymerase Chain Reaction (RT-PCR).
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. The patient has normal organ functions.
7. If the patient is female, she must be of non-childbearing potential, or, if she is of childbearing potential, she must practice adequate contraception for 30 days prior to administration of study treatment, have a negative pregnancy test and continue such precautions during all the study treatment period and for 2 months after completion of the treatment administration series.
8. In the view of the investigator, the patient can and will comply with the requirements of the protocol.

Exclusion Criteria:

1. The patient has at any time received systemic (bio)-chemotherapy.
2. The patient is scheduled to receive any other anticancer treatments than those specified in the protocol, including but not limited to (bio)-chemotherapy, immunomodulating agents and radiotherapy.
3. The patient requires concomitant treatment with systemic corticosteroids, or any other immunosuppressive agents.
4. The patient received any cancer immunotherapeutic containing a MAGE-A3 antigen or any cancer immunotherapeutic for his/her metastatic disease.
5. The patient has received any investigational or non-registered drug or vaccine other than the study medication within the 30 days preceding the first dose of study treatment, or plans to receive such a drug during the study period.
6. The patient has (or has had) previous or concomitant malignancies at other sites, except effectively treated malignancy that is considered by the investigator highly likely to have been cured.
7. History of allergic disease or reactions likely to be exacerbated by any component of the study investigational product.
8. The patient has an autoimmune disease such as, but not limited to, multiple sclerosis, lupus, and inflammatory bowel disease. Patients with vitiligo are not excluded.
9. The patient has a family history of congenital or hereditary immunodeficiency.
10. The patient is known to be positive for the Human Immunodeficiency Virus (HIV).
11. The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent, or to comply with the trial procedures.
12. The patient has concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
13. For female patients: the patient is pregnant or lactating.
14. The patient has an uncontrolled bleeding disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-05-26 (Actual); Primary Completion 2014-11-17 (Actual); Study Completion 2014-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- Belgium (4):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Roeselare
  - GSK Investigational Site, Yvoir
- France (7):
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Villejuif

REFERENCES:
- [Derived] Grob JJ, Mortier L, D'Hondt L, Grange F, Baurain JF, Dreno B, Lebbe C, Robert C, Dompmartin A, Neyns B, Gillet M, Louahed J, Jarnjak S, Lehmann FF. Safety and immunogenicity of MAGE-A3 cancer immunotherapeutic with dacarbazine in patients with MAGE-A3-positive metastatic cutaneous melanoma: an open phase I/II study with a first assessment of a predictive gene signature. ESMO Open. 2017 Nov 14;2(5):e000203. doi: 10.1136/esmoopen-2017-000203. eCollection 2017. PMID 29177094

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the patients and signing informed consent forms.
Groups:
- GSK2132231A GROUP: Patients planned to receive intramuscularly up to 24 doses of GSK2132231A, in 4 cycles.
Period: Overall Study
Arm/Group | GSK2132231A GROUP
Started | 48
Completed | 1
Not Completed | 47
Not completed — Death | 28
Not completed — Ongoing (unknown completion status) | 11
Not completed — Others | 6
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- GSK2132231A GS+ Group: Subset of patients with the pre-specified gene signature, receiving the GSK2132231A product. Gene-signature sub-grouping was based on patients having a potentially predictive gene signature, as assessed at screening.
- GSK2132231A GS- Group: Subset of patients without the pre-specified gene signature, receiving the GSK2132231A product. Gene-signature sub-grouping was based on patients having a potentially predictive gene signature, as assessed at screening.
- GSK2132231A GS Unknown Group: Subset of patients with unknown status as regards GS signature, receiving the GSK2132231A product. Gene-signature sub-grouping was based on patients having a potentially predictive gene signature, as assessed at screening.
- Total: Total of all reporting groups
Arm/Group | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS Unknown Group | Total
Number analyzed (Participants) | 32 | 15 | 1 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.8 (15.4) | 56.1 (18) | 66 (0) | 55.44 (15.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 5 | 0 | 21
  Male | 16 | 10 | 1 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reported With Unsolicited Adverse Events (AEs) That Were Causally Related to Treatment Administration by Maximum Grade.
Description: The assessed AEs were ASCI-related grade 3/4 adverse events according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. An unsolicited AE covers any untoward medical occurrence in a clinical investigation patient temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Related = AE assessed by the investigator as related to the treatment.
Time Frame: Within the 31-day (Days 0-30) post-administration period.
Population: The Total Treated population included all patients who have received at least one dose of the GSK2132231A product.
Measure: Number; unit: Patients
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Patients
  Any event, Grade 3 | 3
  Any event, Grade 4 | 1
  Any Blood and lymphatic system disorders, Grade 3 | 1
  Any Blood and lymphatic system disorders, Grade 4 | 1
  Anaemia, Grade 3 | 0
  Anaemia, Grade 4 | 0
  Lymphopenia, Grade 3 | 0
  Lymphopenia, Grade 4 | 0
  Neutropenia, Grade 3 | 1
  Neutropenia, Grade 4 | 1
  Thrombocytopenia, Grade 3 | 0
  Thrombocytopenia, Grade 4 | 1
  Any Cardiac disorders, Grade 3 | 0
  Any Cardiac disorders, Grade 4 | 0
  Tachycardia, Grade 3 | 0
  Tachycardia, Grade 4 | 0
  Any Gastrointestinal disorders, Grade 3 | 0
  Any Gastrointestinal disorders, Grade 4 | 0
  Constipation, Grade 3 | 0
  Constipation, Grade 4 | 0
  Diarrhoea, Grade 3 | 0
  Diarrhoea, Grade 4 | 0
  Dyspepsia, Grade 3 | 0
  Dyspepsia, Grade 4 | 0
  Nausea, Grade 3 | 0
  Nausea, Grade 4 | 0
  Paraesthesia oral, Grade 3 | 0
  Paraesthesia oral, Grade 4 | 0
  Vomiting, Grade 3 | 0
  Vomiting, Grade 4 | 0
  Any Gen. disord. and adm. site conditions, Grade 3 | 1
  Any Gen. disord. and adm. site conditions, Grade 4 | 0
  Asthenia, Grade 3 | 0
  Asthenia, Grade 4 | 0
  Chills, Grade 3 | 0
  Chills, Grade 4 | 0
  Fatigue, Grade 3 | 0
  Fatigue, Grade 4 | 0
  Influenza like illness, Grade 3 | 0
  Influenza like illness, Grade 4 | 0
  Injection site erythema, Grade 3 | 0
  Injection site erythema, Grade 4 | 0
  Injection site inflammation, Grade 3 | 1
  Injection site inflammation, Grade 4 | 0
  Injection site oedema, Grade 3 | 0
  Injection site oedema, Grade 4 | 0
  Injection site pain, Grade 3 | 0
  Injection site pain, Grade 4 | 0
  Injection site reaction, Grade 3 | 0
  Injection site reaction, Grade 4 | 0
  Mucosal dryness, Grade 3 | 0
  Mucosal dryness, Grade 4 | 0
  Oedema peripheral, Grade 3 | 0
  Oedema peripheral, Grade 4 | 0
  Pyrexia, Grade 3 | 0
  Pyrexia, Grade 4 | 0
  Any Investigations, Grade 3 | 1
  Any Investigations, Grade 4 | 0
  Haemoglobin decreased, Grade 3 | 1
  Haemoglobin decreased, Grade 4 | 0
  Any Metabolism and nutrition disorders, Grade 3 | 0
  Any Metabolism and nutrition disorders, Grade 4 | 0
  Decreased appetite, Grade 3 | 0
  Decreased appetite, Grade 4 | 0
  Any Musculoskeletal and conn. Tiss. Diso., Grade 3 | 0
  Any Musculoskeletal and conn. Tiss. Diso., Grade 4 | 0
  Arthralgia, Grade 3 | 0
  Arthralgia, Grade 4 | 0
  Myalgia, Grade 3 | 0
  Myalgia, Grade 4 | 0
  Pain in extremity, Grade 3 | 0
  Pain in extremity, Grade 4 | 0
  Any Nervous system disorders, Grade 3 | 0
  Any Nervous system disorders, Grade 4 | 0
  Burning sensation, Grade 3 | 0
  Burning sensation, Grade 4 | 0
  Headache, Grade 3 | 0
  Headache, Grade 4 | 0
  Paraesthesia, Grade 3 | 0
  Paraesthesia, Grade 4 | 0
  Presyncope, Grade 3 | 0
  Presyncope, Grade 4 | 0
  Any Psychiatric disorders, Grade 3 | 0
  Any Psychiatric disorders, Grade 4 | 0
  Insomnia, Grade 3 | 0
  Insomnia, Grade 4 | 0
  Any Resp., thoracic and mediastinal. dis., Grade 3 | 0
  Any Resp., thoracic and mediastinal. dis., Grade 4 | 0
  Rhinitis allergic, Grade 3 | 0
  Rhinitis allergic, Grade 4 | 0
  Any Skin and subcutaneous tissue disorder, Grade 3 | 0
  Any Skin and subcutaneous tissue disorder, Grade 4 | 0
  Alopecia, Grade 3 | 0
  Alopecia, Grade 4 | 0
  Eczema, Grade 3 | 0
  Eczema, Grade 4 | 0
  Photosensitivity reaction, Grade 3 | 0
  Photosensitivity reaction, Grade 4 | 0
  Pruritus, Grade 3 | 0
  Pruritus, Grade 4 | 0
  Any Vascular disorders, Grade 3 | 0
  Any Vascular disorders, Grade 4 | 0
  Hypotension, Grade 3 | 0
  Hypotension, Grade 4 | 0

2. Primary Outcome: Number of Patients Reported With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Events which were part of the natural course of the disease under study (i.e., disease progression, recurrence) were captured as part of the clinical activity outcome variables in this study; therefore these did not need to be reported as SAEs. Progression/recurrence of the tumor in a patient was recorded as part of the clinical assessment data collection, and deaths due to progressive disease was recorded on a specific form, but not as an SAE. However, if the investigator considered that there was a causal relationship between treatment or protocol design/procedures and the disease progression/recurrence, then the event was reported as an SAE. Any new primary cancer (non-related to the cancer under study) was reported as an SAE.
Time Frame: During the entire study period, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of the GSK2132231A product.
Measure: Number; unit: Patients
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Patients | 10

3. Primary Outcome: Number of Seroconverted Patients for Melanoma Antigen (Anti-MAGE-A3)
Description: Seroconversion was defined as a concentration of antibodies assessed that was greater than the cut-off value for a patient whose concentration of such antibodies was below the cut-off level before the initiation of treatment. Seroconverted patients were those patients with anti-MAGE-A3 antibody concentrations ≥ 27.
Time Frame: Post Dose 4 at Week 13 (W13).
Population: The Total Treated population included all patients who have received at least one dose of the GSK2132231A product.
Measure: Number; unit: Patients
Arm/Group | GSK2132231A GROUP | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS Unknown Group
Number analyzed (Participants) | 28 | 19 | 8 | 1
Patients | 28 | 19 | 8 | 1

4. Primary Outcome: Anti-MAGE-A3 Antibody Concentrations
Description: Anti-MAGE-A3 antibody concentrations were presented as geometric mean concentrations (GMTs) and expressed in ELISA units per millilitre (EL.U/mL)
Time Frame: Post Dose 4 at Week 13 (W13).
Population: The ATP population for Immunogenecity included all eligible patients, who have received at least the first 4 GSK2132231A doses concomitantly to the standard chemotherapy regimen and provided a valid result for immunogenecity measurement within the 4 weeks following the 4th dose.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK2132231A GROUP | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS Unknown Group
Number analyzed (Participants) | 28 | 19 | 8 | 1
EL.U/mL | 2778.7 [1638.3 to 4712.8] | 2650.8 [1425.5 to 4929.2] | 4046.9 [1206.5 to 13574.7] | 336.0 [NA to NA] — As this analysis was performed on 1 patient, there were no statistics per se, hence no confidence intervals.

5. Primary Outcome: Number of Patients With Treatment Response for Anti-MAGE-A3 Antibodies
Description: Treatment response defined as: For initially seronegative patients: post-administration antibody concentration ≥ 27 EL.U/mL For initially seropositive patients: post-administration antibody concentration ≥ 2 fold the pre-vaccination antibody concentration
Time Frame: Post Dose 4 at Week 13 (W13).
Population: as for outcome 4
Measure: Number; unit: Patients
Arm/Group | GSK2132231A GROUP | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS Unknown Group
Number analyzed (Participants) | 28 | 19 | 8 | 1
Patients | 28 | 19 | 8 | 1

6. Primary Outcome: Concentrations of Antibodies Against Protein D (Anti-PD)
Description: Anti-PD antibody concentrations were presented ad geometric mean concentrations (GMTs) and expressed in ELISA units per millilitre (EL.U/mL).
Time Frame: Post Dose 4 at Week 13 (W13).
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK2132231A GROUP | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS Unknown Group
Number analyzed (Participants) | 28 | 19 | 8 | 1
EL.U/mL | 9979.6 [6470 to 15393] | 10437 [5932.8 to 18361] | 10853.6 [4823.4 to 24422.7] | 2176 [NA to NA] — As the analysis was performed on 1 patient, there were no statistics per se and hence no confidence interval.

7. Primary Outcome: Number of Patients With Treatment Response for Anti-PD
Description: Treatment response defined as: For initially seronegative patients: post-administration antibody concentration ≥ 100 EL.U/mL For initially seropositive patients: post-administration antibody concentration ≥ 2 fold the pre-vaccination antibody concentration
Time Frame: Post Dose 4 at Week 13 (W13).
Population: as for outcome 4
Measure: Number; unit: Patients
Arm/Group | GSK2132231A GROUP | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS Unknown Group
Number analyzed (Participants) | 28 | 19 | 8 | 1
Patients | 28 | 19 | 8 | 1

8. Primary Outcome: Anti-MAGE-A3 Antibody Concentrations (CMI)
Description: Analysis of MAGE-A3 cellular response was not performed and data were not collected..
Time Frame: Post Dose 4 at Week 13 (W13).
Arm/Group | GSK2132231A GROUP | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS Unknown Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Patients With Objective Tumor Response (OR) to MAGE-A3 ASCI Study Treatment
Description: Response assessment was done based on a set of measurable lesions (MLs) identified at baseline as target lesions (TLs), and followed up until disease progression. Up to 5 MLs per organ & 10 in total were identified as TLs and measured at baseline, selected based on size (those with the longest diameter [LD]) and measurability; a sum of LDs for all TLs was calculated and reported as baseline sum LD, which was used to characterize objective tumor response (OR), OR being defined as either complete response (CR) and/or partial response (PR) post MAGE-A3 ASCI treatment. After identification, MLs and TLs were assessed as regards CR and PR definitions per Response Evaluation Criteria in Solid Tumors (RECIST) criteria: CR = Disappearance of all extranodal target lesions. All pathological lymph nodes must have decreased to <10 mm in short axis; PR = At least a 30% decrease in the SLD of target lesions, taking as reference the baseline sum diameters.
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of the GSK2132231A product.
Measure: Number; unit: patients
Arm/Group | GSK2132231A GROUP | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS Unknown Group
Number analyzed (Participants) | 48 | 32 | 15 | 1
patients
  OR | 4 | 4 | 0 | 0
  CR | 1 | 1 | 0 | 0
  PR | 3 | 3 | 0 | 0

10. Secondary Outcome: Number of Patients With Stable Disease (SD) Response to MAGE-A3 ASCI Study Treatment
Description: Assessment was done based on a set of MLs identified at baseline as TLs and NTLs followed up until disease progression. TLs and NTLs were assessed as regards matching or not SD-related definitions, 1) SD definitions per Response Evaluation Criteria in Solid Tumors (RECIST) criteria for TLs >= 20 mm and TLs both >= and < 20 mm: a) for TLs: SD = Neither sufficient shrinkage to qualify as a PR nor sufficient increase to qualify as PD, taking as references the smallest sum LD since treatment start. and b) for NTLs: SD = Persistence of one or more NTL; 2) following below criteria for TLs < 20mm e. a. a) for TLs: PR/SD = Neither sufficient shrinkage to qualify for CR nor sufficient increase, to qualify for PD taking as references the smallest sum LD since treatment start, and b) for NTLs: PR/SD = Persistence of one or more NTL.
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of the GSK2132231A product.
Measure: Number; unit: patients
Arm/Group | GSK2132231A GROUP | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS Unknown Group
Number analyzed (Participants) | 48 | 32 | 15 | 1
patients
  SD | 5 | 4 | 0 | 1
  SD/PR | 0 | 0 | 0 | 0

11. Secondary Outcome: Duration of Stable Disease (SD) Response to MAGE-A3 ASCI Study Treatment
Description: Assessment was done based on a set of MLs identified at baseline as TLs and NTLs followed up until disease progression. Stable disease was defined as follows: 1) In case of target lesions (TL) greater than or equal to (≥) 20 mm: neither sufficient shrinkage to qualify for Partial Response nor sufficient increase to qualify for Progressive Disease, taking as references the sum of Longest Diameter (LD) of TL recorded previously but not necessarily at baseline; 2) In case of TL both less than 20 mm and ≥ 20 mm: Neither sufficient shrinkage to qualify as a PR nor sufficient increase to qualify as PD, taking as references the smallest sum LD since the start of the treatment. The minimal time interval required between 2 measurements for determination of SD was at least 12 weeks.
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of the GSK2132231A product.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS Unknown Group
Number analyzed (Participants) | 6 | 2 | 1
Months | 5.6 [5.3 to 8.3] | 7.7 [7.2 to 8.3] | 5.1 [NA to NA] — The limits for the confidence interval were not available.

12. Secondary Outcome: Number of Patients With Mixed Response (MxR) to MAGE-A3 ASCI Study Treatment
Description: Assessment was done based on a set of MLs identified at baseline as TLs and NTLs followed up until disease progression. MLs were assessed as regards matching below MxR definitions. In case of evaluability per RECIST: a) MxR Type 1= at least (a.l.) 30% decrease in LD in a.l. one TL measured at baseline. Such response occurring in SD/PD status of LD of TL and without appearance of one or more new lesions = SD/PD with TL regression; b) MxR Type 2: appearance of one or more new lesions occurring in SD/PR status of LD of TL, and = SD/PR with new lesion. In case of non-evaluability per RECIST: a) MxR Type 1 = a clear decrease in diameters occurring in a.l. one TL measured at baseline. Such response occurring in SD/PD status of LD of (baseline) TL and without appearance of one or more new lesions = SD/PD with TL regression; b) MxR Type 2 = appearance of one or more new lesions occurring in SD/PR status of LD of TL = SD/PR with new lesion.
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of the GSK2132231A product.
Measure: Number; unit: Patients
Arm/Group | GSK2132231A GROUP | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS Unknown Group
Number analyzed (Participants) | 48 | 32 | 15 | 1
Patients
  MxR: SD/PR with new lesion | 10 | 6 | 4 | 0
  MxR: SD/PD with target lesion regression | 1 [lower limit 0] | 0 | 1 | 0

13. Secondary Outcome: Time to Treatment Failure (TTF), by Gene Signature
Description: TTF was defined as withdrawal from treatment with the MAGE-A3 ASCI study product due to disease progression or death. TTF analysis was performed using the non-parametric Kaplan-Meier method.
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of the GSK2132231A product.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS Unknown Group
Number analyzed (Participants) | 32 | 15 | 1
Months | 2.8 [2.1 to 4.9] | 2.3 [2.1 to 3] | 4.3 [NA to NA] — The limits for the confidence interval were not available.

14. Secondary Outcome: Progression-free Survival (PFS) for the Overall Population
Description: PFS was defined and calculated as the time from first treatment to either the first progression of the disease or the date of death, whichever occurred first. In case a patient went off protocol treatment, the date of first documented progression (if applicable) was to be used as date of progression. Patients still alive with no evidence of disease progression at the time of their last visit or for whom date of first documented progression was not applicable, were censored at the time of the last examination. PFS analysis was performed using the non-parametric Kaplan-Meier method.
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of the GSK2132231A product.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Months | 2.8 [2.8 to 3]

15. Secondary Outcome: Progression-free Survival (PFS) by Gene Signature
Description: as for outcome 14
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of the GSK2132231A product.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | GSK2132231A GROUP | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS Unknown Group
Number analyzed (Participants) | 48 | 32 | 15 | 1
Months | 2.8 [2.8 to 3] | 2.8 [2.8 to 3.4] | 2.8 [2.2 to 3.3] | 5.1 [NA to NA] — The limits for the confidence interval were not available.

16. Secondary Outcome: Progression-free Survival (PFS) After Slow Progressive Disease (SPD) by Gene Signature
Description: PFS after initial SPD was defined and calculated as the time from the time point at which the disease was the most advanced during the treatment to either a new progression of the disease or the date to death, whichever occurred first as another secondary outcome of this study. In that case, the largest diameter during the course of treatment was to be used as reference measurement. This outcome was defined to take into account the delay to induce an active immune response and the strict rules set up in this study to allow pursuing investigational treatment in case of SPD. PFS after SPD analysis was performed using the non-parametric Kaplan-Meier method.
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of the GSK2132231A product.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS Unknown Group
Number analyzed (Participants) | 32 | 15 | 1
Months | 2.8 [2.8 to 5.3] | 2.8 [2.2 to 3.3] | 5.1 [NA to NA] — The limits for the confidence interval were not available.

17. Secondary Outcome: Overall Survival (OS) by Gene Signature
Description: OS was defined as the time from first treatment to the date of death. OS analysis was performed using the non-parametric Kaplan-Meier method. Each patient was censored out at the time of death.
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of the GSK2132231A product.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | GSK2132231A GROUP | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS Unknown Group
Number analyzed (Participants) | 48 | 32 | 15 | 1
Months | 9.4 [5.8 to 15.8] | 11.4 [7.3 to 17.1] | 5.3 [3.3 to 10.5] | 0 [NA to NA] — The limits for the confidence interval were not available.

18. Secondary Outcome: Number of Patients With Abnormal Alanine Aminotransferase (ALT) Values by Maximum Grade
Description: The status of each patient as regards ALT laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0), G1 and G2. CTC grade statuses reported at SE were G0, G1, G2, G3, G4, and Unknown (UNK).
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of the GSK2132231A product.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  ALT - SCR G0; SE G0 | 34
  ALT - SCR G0; SE G1 | 3
  ALT - SCR G0; SE G2 | 1
  ALT - SCR G0; SE G3 | 1
  ALT - SCR G0; SE G4 | 0
  ALT - SCR G0; SE UNK | 1
  ALT - SCR G1; SE G0 | 3
  ALT - SCR G1; SE G1 | 2
  ALT - SCR G1; SE G2 | 1
  ALT - SCR G1; SE G3 | 0
  ALT - SCR G1; SE G4 | 0
  ALT - SCR G1; SE UNK | 1
  ALT - SCR G2; SE G0 | 0
  ALT - SCR G2; SE G1 | 1
  ALT - SCR G2; SE G2 | 0
  ALT - SCR G2; SE G3 | 0
  ALT - SCR G2; SE G4 | 0
  ALT - SCR G2; SE UNK | 0

19. Secondary Outcome: Number of Patients With Abnormal Aspartate Aminotransferase (AST) Values by Maximum Grade
Description: The status of each patient as regards AST laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0) and G1. CTC grade statuses reported at SE were G0, G1, G2, G3, G4, and Unknown (UNK).
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  AST - SCR G0; SE G0 | 36
  AST - SCR G0; SE G1 | 2
  AST - SCR G0; SE G2 | 1
  AST - SCR G0; SE G3 | 0
  AST - SCR G0; SE G4 | 1
  AST - SCR G0; SE UNK | 1
  AST - SCR G1; SE G0 | 2
  AST - SCR G1; SE G1 | 3
  AST - SCR G1; SE G2 | 1
  AST - SCR G1; SE G3 | 0
  AST - SCR G1; SE G4 | 0
  AST - SCR G1; SE UNK | 1

20. Secondary Outcome: Number of Patients With Abnormal Alkaline Phosphatase (ALK) Values by Maximum Grade
Description: The status of each patient as regards ALK laboratory values at baseline (SCR) up to study end(SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0) and G1. CTC grade statuses reported at SE were G0, G1, G2, G3, G4, and Unknown (UNK).
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  ALK - SCR G0; SE G0 | 31
  ALK - SCR G0; SE G1 | 11
  ALK - SCR G0; SE G2 | 0
  ALK - SCR G0; SE G3 | 0
  ALK - SCR G0; SE G4 | 0
  ALK - SCR G0; SE UNK | 1
  ALK - SCR G1; SE G0 | 1
  ALK - SCR G1; SE G1 | 3
  ALK - SCR G1; SE G2 | 0
  ALK - SCR G1; SE G3 | 0
  ALK - SCR G1; SE G4 | 0
  ALK - SCR G1; SE UNK | 1

21. Secondary Outcome: Number of Patients With Abnormal Bilirubine (BIL) Values by Maximum Grade.
Description: The status of each patient as regards BIL laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Unknown (UNK) and Grade 0 (G0). CTC grade statuses reported at SE were G0, G1, G2, G3, G4, and Unknown (UNK).
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  BIL - SCR UNK; SE G0 | 1
  BIL - SCR UNK; SE G1 | 0
  BIL - SCR UNK; SE G2 | 0
  BIL - SCR UNK; SE G3 | 0
  BIL - SCR UNK; SE G4 | 0
  BIL - SCR UNK; SE UNK | 0
  BIL - SCR G0; SE G0 | 39
  BIL - SCR G0; SE G1 | 3
  BIL - SCR G0; SE G2 | 0
  BIL - SCR G0; SE G3 | 0
  BIL - SCR G0; SE G4 | 0
  BIL - SCR G0; SE UNK | 5

22. Secondary Outcome: Number of Patients With Abnormal Creatinine (CREA) Values by Maximum Grade
Description: The status of each patient as regards CREA laboratory values at baseline (SCR) up to study end(SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0). CTC grade statuses reported at SE were G0, G1, G2, G3, G4, and Unknown (UNK).
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  CREA - SCR G0; SE G0 | 40
  CREA - SCR G0; SE G1 | 4
  CREA - SCR G0; SE G2 | 1
  CREA - SCR G0; SE G3 | 0
  CREA - SCR G0; SE G4 | 1
  CREA - SCR G0; SE UNK | 2

23. Secondary Outcome: Number of Patients With Abnormal Gamma-glutamyl Transpeptidase (GGT) Values by Maximum Grade
Description: The status of each patient as regards GGT laboratory values at baseline (SCR) up to study end(SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0), G1 and G3. CTC grade statuses reported at SE were G0, G1, G2, G3, G4, and Unknown (UNK).
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  GGT - SCR G0; SE G0 | 20
  GGT - SCR G0; SE G1 | 11
  GGT - SCR G0; SE G2 | 4
  GGT - SCR G0; SE G3 | 0
  GGT - SCR G0; SE G4 | 0
  GGT - SCR G0; SE UNK | 2
  GGT - SCR G1; SE G0 | 2
  GGT - SCR G1; SE G1 | 2
  GGT - SCR G1; SE G2 | 0
  GGT - SCR G1; SE G3 | 0
  GGT - SCR G1; SE G4 | 0
  GGT - SCR G1; SE UNK | 0
  GGT - SCR G3; SE G0 | 0
  GGT - SCR G3; SE G1 | 0
  GGT - SCR G3; SE G2 | 0
  GGT - SCR G3; SE G3 | 1
  GGT - SCR G3; SE G4 | 0
  GGT - SCR G3; SE UNK | 0

24. Secondary Outcome: Number of Patients With Abnormal Hemoglobin (HGB) Values by Maximum Grade
Description: The status of each patient as regards HGB laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0) and G1. CTC grade statuses reported at SE were G0, G1, G2, G3, G4, and Unknown (UNK).
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  HGB - SCR G0; SE G0 | 22
  HGB - SCR G0; SE G1 | 14
  HGB - SCR G0; SE G2 | 5
  HGB - SCR G0; SE G3 | 1
  HGB - SCR G0; SE G4 | 0
  HGB - SCR G0; SE UNK | 2
  HGB - SCR G1; SE G0 | 2
  HGB - SCR G1; SE G1 | 2
  HGB - SCR G1; SE G2 | 0
  HGB - SCR G1; SE G3 | 0
  HGB - SCR G1; SE G4 | 0
  HGB - SCR G1; SE UNK | 0

25. Secondary Outcome: Number of Patients With Abnormal Hypercalcemia (HCA) Values by Maximum Grade
Description: The status of each patient as regards HCA laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Unknown (UNK), Grade 0 (G0) and G1. CTC grade statuses reported at SE were G0, G1, G2, G3, G4, and Unknown (UNK).
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  HCA - SCR UNK; SE G0 | 2
  HCA - SCR UNK; SE G1 | 1
  HCA - SCR UNK; SE G2 | 0
  HCA - SCR UNK; SE G3 | 0
  HCA - SCR UNK; SE G4 | 0
  HCA - SCR UNK; SE UNK | 0
  HCA - SCR G0; SE G0 | 37
  HCA - SCR G0; SE G1 | 0
  HCA - SCR G0; SE G2 | 0
  HCA - SCR G0; SE G3 | 0
  HCA - SCR G0; SE G4 | 0
  HCA - SCR G0; SE UNK | 6
  HCA - SCR G1; SE G1 | 1
  HCA - SCR G1; SE G2 | 1
  HCA - SCR G1; SE G3 | 0
  HCA - SCR G1; SE G4 | 0
  HCA - SCR G1; SE UNK | 0

26. Secondary Outcome: Number of Patients With Abnormal Hyperkalemia (HKA) Values by Maximum Grade
Description: The status of each patient as regards HKA laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0), G1 and G2. CTC grade statuses reported at SE were G0, G1, G2, G3, G4, and Unknown (UNK).
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  HKA - SCR G0; SE G0 | 42
  HKA - SCR G0; SE G1 | 2
  HKA - SCR G0; SE G2 | 0
  HKA - SCR G0; SE G3 | 0
  HKA - SCR G0; SE G4 | 0
  HKA - SCR G0; SE UNK | 1
  HKA - SCR G1; SE G0 | 1
  HKA - SCR G1; SE G1 | 0
  HKA - SCR G1; SE G2 | 0
  HKA - SCR G1; SE G3 | 0
  HKA - SCR G1; SE G4 | 0
  HKA - SCR G1; SE UNK | 1
  HKA - SCR G2; SE G0 | 1
  HKA - SCR G2; SE G1 | 0
  HKA - SCR G2; SE G2 | 0
  HKA - SCR G2; SE G3 | 0
  HKA - SCR G2; SE G4 | 0
  HKA - SCR G2; SE UNK | 0

27. Secondary Outcome: Number of Patients With Abnormal Hypernatremia (HNA) Values by Maximum Grade
Description: The status of each patient as regards HNA laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0) and G1. CTC grade statuses reported at SE were G0, G1, G2, G3, G4, and Unknown (UNK).
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  HNA - SCR G0; SE G0 | 44
  HNA - SCR G0; SE G1 | 0
  HNA - SCR G0; SE G2 | 0
  HNA - SCR G0; SE G3 | 0
  HNA - SCR G0; SE G4 | 0
  HNA - SCR G0; SE UNK | 2
  HNA - SCR G1; SE G0 | 2
  HNA - SCR G1; SE G1 | 0
  HNA - SCR G1; SE G2 | 0
  HNA - SCR G1; SE G3 | 0
  HNA - SCR G1; SE G4 | 0
  HNA - SCR G1; SE UNK | 0

28. Secondary Outcome: Number of Patients With Abnormal Hypoalbuminemia(hAL) Values by Maximum Grade
Description: The status of each patient as regards hAL laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Unknown (UNK), Grade 0 (G0) and G1. CTC grade statuses reported at SE were G0, G1, G2, G3, G4, and Unknown (UNK).
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  hAL - SCR UNK; SE G0 | 1
  hAL - SCR UNK; SE G1 | 0
  hAL - SCR UNK; SE G2 | 1
  hAL - SCR UNK; SE G3 | 0
  hAL - SCR UNK; SE G4 | 0
  hAL - SCR UNK; SE UNK | 1
  hAL - SCR G0; SE G0 | 26
  hAL - SCR G0; SE G1 | 4
  hAL - SCR G0; SE G2 | 2
  hAL - SCR G0; SE G3 | 0
  hAL - SCR G0; SE G4 | 0
  hAL - SCR G0; SE UNK | 4
  hAL - SCR G1; SE G1 | 4
  hAL - SCR G1; SE G2 | 3
  hAL - SCR G1; SE G3 | 0
  hAL - SCR G1; SE G4 | 0
  hAL - SCR G1; SE UNK | 2

29. Secondary Outcome: Number of Patients With Abnormal Hypocalcemia(hCA) Values by Maximum Grade
Description: as for outcome 25
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  hCA - SCR UNK; SE G0 | 1
  hCA - SCR UNK; SE G1 | 1
  hCA - SCR UNK; SE G2 | 0
  hCA - SCR UNK; SE G3 | 0
  hCA - SCR UNK; SE G4 | 1
  hCA - SCR UNK; SE UNK | 0
  hCA - SCR G0; SE G0 | 27
  hCA - SCR G0; SE G1 | 7
  hCA - SCR G0; SE G2 | 0
  hCA - SCR G0; SE G3 | 0
  hCA - SCR G0; SE G4 | 0
  hCA - SCR G0; SE UNK | 5
  hCA - SCR G1; SE G0 | 0
  hCA - SCR G1; SE G1 | 5
  hCA - SCR G1; SE G2 | 0
  hCA - SCR G1; SE G3 | 0
  hCA - SCR G1; SE G4 | 0
  hCA - SCR G1; SE UNK | 1

30. Secondary Outcome: Number of Patients With Abnormal Hypokalemia (hKA) Values by Maximum Grade
Description: The status of each patient as regards hKA laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0) and G1. CTC grade statuses reported at SE were G0, G1, G2, G3, G4, and Unknown (UNK).
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  hKA - SCR G0; SE G0 | 42
  hKA - SCR G0; SE G1 | 1
  hKA - SCR G0; SE G2 | 0
  hKA - SCR G0; SE G3 | 0
  hKA - SCR G0; SE G4 | 0
  hKA - SCR G0; SE UNK | 1
  hKA - SCR G1; SE G0 | 3
  hKA - SCR G1; SE G1 | 0
  hKA - SCR G1; SE G2 | 0
  hKA - SCR G1; SE G3 | 0
  hKA - SCR G1; SE G4 | 0
  hKA - SCR G1; SE UNK | 1

31. Secondary Outcome: Number of Patients With Abnormal Hyponatremia (hNA) Values by Maximum Grade
Description: as for outcome 27
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  hNA - SCR G0; SE G0 | 33
  hNA - SCR G0; SE G1 | 10
  hNA - SCR G0; SE G2 | 0
  hNA - SCR G0; SE G3 | 1
  hNA - SCR G0; SE G4 | 0
  hNA - SCR G0; SE UNK | 2
  hNA - SCR G1; SE G0 | 1
  hNA - SCR G1; SE G1 | 1
  hNA - SCR G1; SE G2 | 0
  hNA - SCR G1; SE G3 | 0
  hNA - SCR G1; SE G4 | 0
  hNA - SCR G1; SE UNK | 0

32. Secondary Outcome: Number of Patients With Abnormal Leukocytes (LEU) Values by Maximum Grade
Description: The status of each patient as regards LEU laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0) and G1. CTC grade statuses reported at SE were G0, G1, G2, G3, G4, and Unknown (UNK).
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  LEU - SCR G0; SE G0 | 37
  LEU - SCR G0; SE G1 | 6
  LEU - SCR G0; SE G2 | 0
  LEU - SCR G0; SE G3 | 1
  LEU - SCR G0; SE G4 | 0
  LEU - SCR G0; SE UNK | 2
  LEU - SCR G1; SE G0 | 0
  LEU - SCR G1; SE G1 | 1
  LEU - SCR G1; SE G2 | 1
  LEU - SCR G1; SE G3 | 0
  LEU - SCR G1; SE G4 | 0
  LEU - SCR G1; SE UNK | 0

33. Secondary Outcome: Number of Patients With Abnormal Lymphopenia (LYM) Values by Maximum Grade
Description: The status of each patient as regards LYM laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0) and G1. CTC grade statuses reported at SE were G0, G1, G2, G3, G4, and Unknown (UNK).
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  LYM - SCR G0; SE G0 | 18
  LYM - SCR G0; SE G1 | 13
  LYM - SCR G0; SE G2 | 6
  LYM - SCR G0; SE G3 | 0
  LYM - SCR G0; SE G4 | 0
  LYM - SCR G0; SE UNK | 2
  LYM - SCR G1; SE G0 | 2
  LYM - SCR G1; SE G1 | 4
  LYM - SCR G1; SE G2 | 3
  LYM - SCR G1; SE G3 | 0
  LYM - SCR G1; SE G4 | 0
  LYM - SCR G1; SE UNK | 0

34. Secondary Outcome: Number of Patients With Abnormal Neutrophils (NEU) Values by Maximum Grade
Description: The status of each patient as regards NEU laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0). CTC grade statuses reported at SE were G0, G1, G2, G3, G4, and Unknown (UNK).
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  NEU - SCR G0; SE G0 | 39
  NEU - SCR G0; SE G1 | 4
  NEU - SCR G0; SE G2 | 1
  NEU - SCR G0; SE G3 | 2
  NEU - SCR G0; SE G4 | 0
  NEU - SCR G0; SE UNK | 2

35. Secondary Outcome: Number of Patients With Abnormal Partial Thromboplastin Time (PTT) Values by Maximum Grade
Description: The status of each patient as regards PTT laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0) and G1. CTC grade statuses reported at SE were G0, G1, G2, G3, G4, and Unknown (UNK).
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  PTT - SCR G0; SE G0 | 35
  PTT - SCR G0; SE G1 | 3
  PTT - SCR G0; SE G2 | 0
  PTT - SCR G0; SE G3 | 1
  PTT - SCR G0; SE G4 | 0
  PTT - SCR G0; SE UNK | 7
  PTT - SCR G1; SE G0 | 0
  PTT - SCR G1; SE G1 | 1
  PTT - SCR G1; SE G2 | 0
  PTT - SCR G1; SE G3 | 1
  PTT - SCR G1; SE G4 | 0
  PTT - SCR G1; SE UNK | 0

36. Secondary Outcome: Number of Patients With Abnormal Platelets(PLT) Values by Maximum Grade
Description: The status of each patient as regards PLT laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0) and G1. CTC grade statuses reported at SE were G0, G1, G2, G3, G4, and Unknown (UNK).
Time Frame: During the entire study, up to 5 years
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  PLT - SCR G0; SE G0 | 39
  PLT - SCR G0; SE G1 | 5
  PLT - SCR G0; SE G2 | 1
  PLT - SCR G0; SE G3 | 0
  PLT - SCR G0; SE G4 | 0
  PLT - SCR G0; SE UNK | 2
  PLT - SCR G1; SE G0 | 1
  PLT - SCR G1; SE G1 | 0
  PLT - SCR G1; SE G2 | 0
  PLT - SCR G1; SE G3 | 0
  PLT - SCR G1; SE G4 | 0
  PLT - SCR G1; SE UNK | 0

37. Secondary Outcome: Number of Patients With Any Adverse Events (AEs) and With AEs by Maximum Grade
Description: An AE was any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs reported are here below tabulated irrespective of grade (any), as well as graded by maximum grade reported according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. Maximum grade reported and tabulated were Grade 1 (G1), G2, G3, G4 and G5.
Time Frame: Within the 31-day follow-up period post treatment administration.
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  Patients with any AEs | 48
  Patients with G1 AEs | 14
  Patients with G2 AEs | 19
  Patients with G3 AEs | 12
  Patients with G4 AEs | 3
  Patients with G5 AEs | 0

38. Secondary Outcome: Number of Patients With Any Serious Adverse Events (SAEs) and With AEs by Maximum Grade
Description: SAEs include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a patient, is a Grade 4 AE according to the CTCAE, version3.0. Events which were part of the natural course of the disease under study were captured as part of the clinical activity outcome variables in this study; therefore did not need to be reported as SAEs. Progression/recurrence of the tumor was recorded as part of the clinical assessment data collection, and deaths due to progressive disease was recorded on a specific form, but not as an SAE. SAEs reported are here below tabulated irrespective of grade (any), as well as graded by maximum grade reported according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. Maximum grade reported and tabulated were Grade 1 (G1), G2, G3, G4 and G5.
Time Frame: Within the 31-day follow-up period post treatment administration.
Population: The Total Treated population included all patients who have received at least one dose of GSK2132231A.
Measure: Number; unit: Subjects
Arm/Group | GSK2132231A GROUP
Number analyzed (Participants) | 48
Subjects
  Patients with any SAEs | 10
  Patients with G1 SAEs | 1
  Patients with G2 SAEs | 2
  Patients with G3 SAEs | 5
  Patients with G4 SAEs | 2
  Patients with G5 SAEs | 0

ADVERSE EVENTS:
Time Frame: SAEs: From screening (SCR) up to study end; AEs: Within the 31-day follow-up period post treatment administration, up to study end.
Description: The occurrence of reported AEs (all/related) was not available and is encoded as equal to the number of subjects affected.
Arm/Group | GSK2132231A GROUP
Serious Adverse Events (participants affected / at risk) | 10/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2132231A GROUP (N=48)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Asthenia (General disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2132231A GROUP (N=48)
Asthenia (General disorders) | 25 (25)
Injection site pain (General disorders) | 18 (18)
Pyrexia (General disorders) | 14 (14)
Injection site reaction (General disorders) | 9 (9)
Influenza like illness (General disorders) | 9 (9)
Fatigue (General disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 22 (22)
Constipation (Gastrointestinal disorders) | 14 (14)
Vomiting (Gastrointestinal disorders) | 13 (13)
Decreased appetite (Metabolism and nutrition disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.